CLINICAL TRIAL: NCT05051878
Title: Effect of T-scan Occlusal Analysis and Adjustment vs Articulating Paper on Stresses Transmitted to Single Mandibular Implant Supported Prosthesis
Brief Title: Effect of T-scan Occlusal Analysis and Adjustment vs Articulating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: OCCLUSAL EVALUATION
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Occlusion
Keywords: t-scan; occlusal analysis; implant supported prosthesis
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- articulating paper occlusal adjustment (Experimental): occlusal adjustments of implant supported prosthesis according to articulating paper occlusal analysis
  Interventions: Other: articulating paper
- T-scan occlusal analysis (Experimental): occlusal adjustments of implant supported prosthesis according to T-scan occlusal analysis
  Interventions: Device: T-scan

INTERVENTIONS:
Device: T-scan — occlusal analysis T-scan
  Arms: T-scan occlusal analysis
Other: articulating paper — articulating paper occlusal analysis
  Arms: articulating paper occlusal adjustment

SUMMARY:
The aim of this study is to compare two different methods for occlusal analysis of implant - supported prosthesis (T-scan and conventional method with articulating papers) regarding the stresses transmitted to the implants.

DETAILED DESCRIPTION:
Four implants will be inserted, two implants in canine regions and two implants in lower second premolar regions.

After 3 months, two identical overdentures will be constructed for the patient on implants.

The occlusion of each one of the two identical prostheses will be adjusted intraorally but according to different occlusal analysis:

* Group (A) : occlusal adjustments for the overdenture will be done according to articulating paper analysis.
* Group (B) :- occlusal adjustments for the overdenture will be done according to T-scan analysis.

The two prostheses will be retained on dummy implants on acrylic cast and will be loaded under chewing simulator.

The strain developed around the dummy implants will be measured. The data will be recorded manually then will be transferred into digital form. The obtained data will be recorded, tabulated and statistically analyzed using the appropriate tests for comparison within each group.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 55-65.
* Radiographic examination should reveal bone height more than 10 mm and crestal bone width not less than 5 mm of the inter-foraminal region.
* Residual bone and mucosa should be free from any pathological signs, bony undercuts, or neoplasia.
* Adequate salivary flow.
* Adequate mouth opening.
* Adequate inter-arch space.

Exclusion Criteria:

* Systemic diseases affecting metabolism of bone e.g uncontrolled diabetes, bone diseases, hyperparathyroidism and renal disease.
* Severe blood diseases (hemophilia etc.).
* Severe vascular heart disease.
* Liver Problems.
* Cerebral infarction .
* Severe immunodeficiency.
* Patients who are undergoing strong chemotherapy.
* Excessive alcohol consumption.
* Severe neuropsychiatric disease, mental disability, and narcotic drug addict
* Uncooperative patients

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
stresses around implants | baseline
  stresses transmitted around implants supporting the prosthesis by stain gauge

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alafandy, professor, Study Director — oral & maxillofacial prosthodontics Faculty of Dentistry Ain-shams University; Ahmed Osama, professor, Study Director — oral & maxillofacial prosthodontics Faculty of Dentistry Ain-shams University; Omar ELsadat, lecturer, Study Director — oral & maxillofacial prosthodontics Faculty of Dentistry Ain-shams University
Locations (1):
- Faculty of dentistry, Ain Shams University, Cairo, Egypt